CLINICAL TRIAL: NCT01441414
Title: A PHASE II TRIAL OF PF-04856884 (CVX-060), A SELECTIVE ANGIOPOIETIN-2 (ANG-2) INHIBITOR IN COMBINATION WITH AG-013736 (AXITINIB) IN PATIENTS WITH PREVIOUSLY TREATED METASTATIC RENAL CELL CARCINOMA
Brief Title: PF-04856884 (CVX-060) In Combination With Axitinib In Patients With Previously Treated Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: B1131004; 2011-002190-33 (EudraCT Number)
Record Dates: First submitted 2011-08-26; First posted 2011-09-27 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: CVX-060; PF-04856884; AG-013736; axitinib; mRCC; metastatic renal cell cancer; second line; anti-angiogenic; Ang-2
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): PF-04856884 in combination with AG-013736
  Interventions: Biological: PF-04856884; Drug: Axitinib (AG-013736)
- ARM B (Active Comparator): AG-013736 alone
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Biological: PF-04856884 — 15 mg/kg/week intravenously [IV] until toxicity or disease progression
  Arms: ARM A
Drug: Axitinib (AG-013736) — 5 mg PO BID
  Arms: ARM A
Drug: Axitinib (AG-013736) — 5 mg PO BID
  Arms: ARM B

SUMMARY:
To evaluate the combination of PF-04856884 (CVX-060) in combination with Axitinib (AG-013736) in patients that have received one prior systemic regimen for metastatic renal cell carcinoma (mRCC) vs. axitinib alone.

DETAILED DESCRIPTION:
The study was prematurely discontinued on 06Nov2012 due to tolerability findings in patients treated in Part I of the study that have prompted the Sponsor to re-evaluate the strategic development of the program. An unexpected frequency of arterial thrombotic events (ATEs) and venous thrombotic events (VTEs) were reported in patients treated in Part I.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients with histologically or cytologically confirmed renal cell cancer (RCC) with a component of clear cell subtype and evidence of metastasis
* Evidence of unidimensionally measurable disease
* Prior therapy: Part I: Having received 1 to 3 prior systemic regimens for treatment of mRCC
* Part II: Evidence of disease progression following 1 prior regimen administered as 1st line therapy for mRCC. The prior regimen must have contained one of the following: VEGFR2 tyrosine kinase inhibitor (TKI) or other anti VEGF [Vascular Endothelial Growth Factor] compounds, such as bevacizumab
* adequate bone marrow, liver and renal function

Exclusion Criteria:

Part I:

* Intolerant to prior AG 013736 therapy or prior treatment with compounds which contain the core platform antibody as PF 04856884

Part II:

* Prior AG 013736 therapy, more than one systemic first-line regimen for the treatment of mRCC and prior treatment with compounds which contain the core platform antibody as PF 04856884
* major surgery <4 weeks or radiation therapy <2 weeks prior to start of therapy
* clinically significant gastrointestinal abnormalities
* current use or anticipated need for drugs that are known potent CYP3A4 inhibitors and drugs that are known CYP3A4 or CYP1A2 inducers
* history of bleeding diathesis or coagulopathy
* Grade 3 or greater hemorrhage from any cause <4 weeks prior to screening;
* hemoptysis >½ teaspoon of blood per day within 2 weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11-21 (Actual); Primary Completion 2014-03-27 (Actual); Study Completion 2014-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- United States (22):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Arizona Oncology Associates, PC-HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Centennial, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Regional Cancer Care-Durham, Durham, North Carolina
  - Texas Oncology-Tyler, Tyler, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Masarykuv onkologicky ustav, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1131004&StudyName=PF-04856884%20%28CVX-060%29%20In%20Combination%20With%20Axitinib%20In%20Patients%20With%20Previously%20Treated%20Metastatic%20Renal%20Cell%20Carcinoma

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, open-label study consisted of a safety lead in stage (Part I) followed by a randomized Phase 2 stage (Part II). A total of 18 participants were screened and assigned to treatment in Part I, with 3 participants completing Part I of the study. At the completion of Part I, all 18 participants had discontinued combined treatment.
Pre-assignment Details: During Part I, 3 to 4 participants were initially treated with the study drug combination in 28-day cycles. If no participants experienced Cycle 1 dose limiting toxicities (DLTs), another 6 to 9 participants were treated at this dose level. Part II of the study was to be initiated if Cycle 1 DLTs were observed in <33% in at least 12 participants.
Groups:
- PF-04856884 + AG-013736: Participants in Part I received PF-04856884 15 mg/kg/week and AG-013736 5 mg twice a day. Following the decision of 06 November 2012 not to continue with Part II of the study, any participant remaining in Part I continued to receive PF-04856884 at a reduced dose of 10 mg/kg/week in combination with AG-013736 (5 mg twice a week) or AG-013736 alone (5 mg twice a week).
Period: Overall Study
Arm/Group | PF-04856884 + AG-013736
Started | 18
Completed | 3
Not Completed | 15
Not completed — Participant died | 9
Not completed — Other reasons | 3
Not completed — Study terminated by sponsor | 2
Not completed — Subject refused further follow-up | 1

BASELINE CHARACTERISTICS:
Population: The full analysis (FA) set was the primary population for evaluating all safety and efficacy endpoints per the treatment randomization as well as participant characteristics.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (AEs) in Part I (Reported in ≥2 of the Participants Overall).
Description: Incidence and severity of all treatment-emergent AEs (TEAEs) of both all-causality and treatment-related by preferred term (PT) categorized according to Common Terminology Criteria for Adverse Events (CTCAE) grades reported in ≥2 participants overall (CTCAE Grades 3, 4 and 5, combined) for any PT are presented. Participants who are included under all-causality TEAE PT are coded as NA if they appear for the same PT under treatment-related TEAE below.
  Participants in Part I received PF-04856884 15 mg/kg/week and AG-013736 5 mg twice daily. Following the decision on 06 November 2012 not to continue with Part II of the study, any participant remaining in Part I continued to receive PF-04856884 at a reduced dose of 10 mg/kg/week in combination with AG-013736 (5 mg twice a week) or AG-013736 alone (5 mg twice a week).
Time Frame: 4 months
Population: The FA set was the primary population for evaluating all safety and efficacy endpoints per the treatment randomization as well as participant characteristics.
Measure: Number; unit: participants
Groups:
- All-causality CTCAE Grade 3: Incidence and severity of all-causality CTCAE Grade 3 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- All-causality CTCAE Grade 4: Incidence and severity of all-causality CTCAE Grade 4 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- All-causality CTCAE Grade 5: Incidence and severity of all-causality CTCAE Grade 5 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- Treatment-related CTCAE Grade 3: Incidence and severity of treatment-related CTCAE Grade 3 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- Treatment-related CTCAE Grade 4: Incidence and severity of treatment-related CTCAE Grade 4 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- Treatment-related CTCAE Grade 5: Incidence and severity of treatment-related CTCAE Grade 5 TEAEs are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- All-causality Overall: Incidence and severity of all-causality CTCAE Grades 3, 4, and 5 are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
- Treatment-related Overall: Incidence and severity of treatment-related CTCAE Grades 3,4, and 5 are presented. Participants with multiple occurrences of an AE within a category were counted once within the category.
Arm/Group | All-causality CTCAE Grade 3 | All-causality CTCAE Grade 4 | All-causality CTCAE Grade 5 | Treatment-related CTCAE Grade 3 | Treatment-related CTCAE Grade 4 | Treatment-related CTCAE Grade 5 | All-causality Overall | Treatment-related Overall
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18 | 18 | 18
participants
  Anaemia | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
  Leukocytosis | 2 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Pericardial effusion | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2
  Hyperthyroidism | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Hypothyroidism | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE
  Vision blurred | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE
  Abdominal pain | 1 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Constipation | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2
  Diarrhoea | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 9
  Dry mouth | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 3 | NA — participant appears for the same preferred term under all-causality TEAE.
  Gastritis | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Nausea | 1 | 0 | 0 | 1 | 0 | 0 | 11 | 7
  Oral pain | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Stomatitis | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Toothache | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Vomiting | 1 | 0 | 0 | 1 | 0 | 0 | 10 | 6
  Asthenia | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
  Fatigue | 5 | 0 | 0 | 4 | 0 | 0 | 11 | 8
  Oedema peripheral | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE.
  Pneumonia | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Upper respiratory tract infection | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Urinary tract infection | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 3 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Blood creatinine increased | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 3 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Weight decreased | 2 | 0 | 0 | 1 | 0 | 0 | 4 | 4
  Decreased appetite | 1 | 0 | 0 | 1 | 0 | 0 | 12 | 11
  Dehydration | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
  Hypercalcaemia | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Hypokalaemia | 1 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Hyponatraemia | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Hypovolaemia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Arthralgia | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 3 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Back pain | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 5 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Muscle spasms | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Muscular weakness | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Myalgia | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Cerebrovascular accident | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2
  Dizziness | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 4 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Headache | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 2
  Migraine | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2
  Neuropathy peripheral | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Depression | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 3 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Insomnia | 1 | 0 | 0 | 1 | 0 | 0 | 7 | 2
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Cough | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 7 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Dysphonia | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5
  Dyspnoea | 1 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 6 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Hypoxia | 1 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 2 | NA — participant appears for the same preferred term under all-causality TEAE.
  Pleural effusion | 1 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 3 | NA — participant appears for the same preferred term under all-causality TEAE.
  Pulmonary embolism | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2
  Night sweats | 0 | 0 | 0 | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | NA — less than 2 participants per preferred term for treatment-related TEAE | 2 | NA — less than 2 participants per preferred term for treatment-related TEAE
  Palmar-plantar erythrodysaesthesia | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Hot flush | 0 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 3 | NA — participant appears for the same preferred term under all-causality TEAE.
  Hypertension | 5 | 0 | 0 | 4 | 0 | 0 | 10 | 9
  Hypotension | 1 | 0 | 0 | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | NA — participant appears for the same preferred term under all-causality TEAE. | 4 | NA — participant appears for the same preferred term under all-causality TEAE.

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Part I
Description: Incidence and severity of all-causality serious adverse events (SAEs) are presented by PT categorized according to Common Terminology Criteria for Adverse Events (CTCAE) grades. Participants in Part I received PF-04856884 15 mg/kg/week and AG-013736 5 mg twice daily. Following the decision on 06 November 2012 not to continue with Part II of the study, any participant remaining in Part I continued to receive PF-04856884 at a reduced dose of 10 mg/kg/week in combination with AG-013736 (5 mg twice a week) or AG-013736 alone (5 mg twice a week). Participants with treatment-related TEAE are coded as NA if they appear for the same preferred term under all-causality TEAE.
Time Frame: 4 months
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- All-causality CTCAE Grade 2: Number of participants who had serious TEAEs (all-causality) of CTCAE Grade 2 TEAEs are presented
- All-causality CTCAE Grade 3: Number of participants who had serious TEAEs (all-causality) of CTCAE Grade 3 TEAEs are presented
- All-causality CTCAE Grade 4: Number of participants who had serious TEAEs (all-causality) of CTCAE Grade 4 TEAEs are presented
- All-causality CTCAE Grade 5: Number of participants who had serious TEAEs (all-causality) of CTCAE Grade 5 TEAEs are presented
Arm/Group | All-causality CTCAE Grade 2 | All-causality CTCAE Grade 3 | All-causality CTCAE Grade 4 | All-causality CTCAE Grade 5
Number analyzed (Participants) | 18 | 18 | 18 | 18
participants
  Pneumonia | 1 | 1 | 0 | 0
  Pleural effusion | 1 | 1 | 0 | 0
  Ileus | 1 | 0 | 0 | 0
  Abdominal pain | 0 | 1 | 0 | 0
  Ascites | 1 | 0 | 0 | 0
  Lung infection | 0 | 1 | 0 | 0
  Back pain | 0 | 1 | 0 | 0
  Musculoskeletal chest pain | 0 | 1 | 0 | 0
  Convulsion | 1 | 0 | 0 | 0
  Embolism | 1 | 0 | 0 | 0
  Hyponatraemia | 0 | 1 | 0 | 0
  Dyspnoea | 0 | 1 | 0 | 0
  Hypotension | 0 | 1 | 0 | 0
  Cerebrovascular accident | 0 | 1 | 1 | 0
  Migraine | 0 | 1 | 0 | 0
  Meningioma | 0 | 1 | 0 | 0
  Hypovolaemia | 1 | 0 | 0 | 0
  Pulmonary embolism | 0 | 1 | 1 | 0
  Pericardial effusion | 0 | 0 | 1 | 0
  Gastrointestinal disorder | 0 | 0 | 0 | 1
  Chest discomfort | 0 | 1 | 0 | 0
  Hypertension | 0 | 1 | 0 | 0

3. Primary Outcome: Progression Free Survival (PFS) in Adult Participants With Previously Treated Metastatic Renal Cell Cancer (mRCC) in Part II
Description: PFS is defined as the time (in days) from date of randomization to first documentation of investigator assessed tumor progression or death, whichever comes first. Progression free survival was to be calculated as (first event date - the date of randomization +1).
Time Frame: 3 years
Population: The primary efficacy endpoint of estimating median PFS in Part II was not assessed due to early termination of the study.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Non-serious AEs and SAEs
Description: Incidence and severity of all-causality AEs and SAEs to be presented by PT categorized according to Common Terminology Criteria for Adverse Events (CTCAE) grades. Participants in Part I received PF-04856884 15 mg/kg/week and AG-013736 5 mg twice daily. Following the decision on 06 November 2012 not to continue with Part II of the study, any participant remaining in Part I continued to receive PF-04856884 at a reduced dose of 10 mg/kg/week in combination with AG-013736 (5 mg twice a week) or AG-013736 alone (5 mg twice a week).
Time Frame: 3 years
Population: This endpoint was not assessed due to the early termination of the study.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Response Rate (ORR) in Metastatic Renal Cell Cancer (mRCC) Patients Treated With PF-04856884 in Combination With AG-013736 vs. AG-013736 Alone.
Description: ORR is defined as the proportion of participants with confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST), relative to all randomized participants as defined in the FA Set. Confirmed responses are those that persist on repeat imaging study ≥ 4 weeks after initial documentation of response. Participants who do not have on-study radiographic tumor evaluation or who die, progress, or drop out for any reason prior to reaching a CR or PR will be counted as non-responders (NR) in the assessment of ORR.
Time Frame: 4 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
Percentage of participants
  Complete response (CR) | 0
  Partial response (PR) | 11.1
  ORR (CR + PR) | 11.1

6. Secondary Outcome: Duration of Response (DR) in Metastatic Renal Cell Cancer (mRCC) Patients Treated With PF-04856884 in Combination With AG-013736 vs. AG-013736 Alone
Description: DR is defined as the time from the first documentation of objective tumor response (CR or PR) that is subsequently confirmed to the first documentation of tumor progression or to death due to cancer. Duration of tumor response was to be calculated as (the end date for DR - first CR or PR that is subsequently confirmed +1).
Time Frame: 3 years
Population: This endpoint was not assessed due to the early termination of the study.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 0

7. Secondary Outcome: Tmax (Time When Maximum Serum PF-04856884 Concentration Was Reached)
Description: Pharmacokinetic parameter, Tmax (Time when maximum serum PF-04856884 concentration was reached) was done using non-compartmental methods.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 192, 360, 361, 362, 365, 367 hours post dose and end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
hr
  CYCLE1/DAY1 | 2.000 (1.6450)
  CYCLE1/DAY22 | 3.000 (2.1122)

8. Secondary Outcome: Cmax (Observed Peak Serum PF-04856884 Concentration)
Description: Pharmacokinetic parameter Cmax (observed peak PF-04856884 serum concentration) was estimated using noncompartmental methods.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 192, 360, 361, 362, 365, 367 hours post dose and end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
ng/mL
  CYCLE1/DAY1 | 337100 (76245)
  CYCLE1/DAY22 | 531400 (154780)

9. Secondary Outcome: Cmin (Trough PF-04856884 Serum Concentration)
Description: Pharmacokinetic parameter Cmin (trough PF-04856884 serum concentration) was estimated using noncompartmental methods.
Time Frame: Pre-dose, 1, 2, 4, 6, 8, 192, 360, 361, 362, 365, 367 hours post dose and end of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
ng/mL
  CYCLE1/DAY1 | 932.7 (3499.1)
  CYCLE1/DAY22 | 168900 (84507)

10. Secondary Outcome: Number of Anti-drug Antibodies (ADA) Samples Confirmed Positive
Description: Detection of neutralizing anti-PF-04856884 antibodies was based on the ability of anti-PF-04856884 neutralizing antibodies to bind to Tag-PF-04856884.
Time Frame: 0 and 360 hours post dose and end of study
Population: as for outcome 1
Measure: Number; unit: ADA samples
Units Other Than Participants: ADA samples
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 18
Number analyzed (ADA samples) | 91
ADA samples | 8

11. Secondary Outcome: Progression Free Survival (PFS) in Adult Participants With Previously Treated Metastatic Renal Cell Cancer (mRCC) as Measured by an Independent Radiological Assessment
Description: PFS is defined as the time (in days) from date of randomization to first documentation of investigator assessed tumor progression or death, whichever comes first. PFS was to be calculated as (first event date - the date of randomization +1).
Time Frame: 3 years
Population: This endpoint of estimating median PFS was not assessed due to early termination of the study.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 0

12. Secondary Outcome: Overall Survival (OS) at 2 Years
Description: OS is defined as the time from the first dose date to date of death. For participants not expiring, their survival times will be censored at the last date they are known to be alive, or 2 year whichever is earlier. The 2-year OS rate will be estimated from a time-to event analysis of OS.
Time Frame: 5 years
Population: This endpoint was not assessed due to the early termination of the study.
Arm/Group | PF-04856884 + AG-013736
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From the day the first dose of the investigational product was administered up to 1 year.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04856884 + AG-013736
Serious Adverse Events (participants affected / at risk) | 12/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04856884 + AG-013736 (N=18)
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Embolism (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04856884 + AG-013736 (N=18)
Anaemia (Blood and lymphatic system disorders) | 4
Leukocytosis (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypothyroidism (Endocrine disorders) | 2
Eye pain (Eye disorders) | 1
Vision blurred (Eye disorders) | 3
Visual impairment (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 3
Eructation (Gastrointestinal disorders) | 1
Faecal incontinence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 11
Oral pain (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 11
Inflammation (General disorders) | 1
Localised oedema (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cyst (Hepatobiliary disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Candida infection (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 3
Procedural pain (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 3
Blood thyroid stimulating hormone increased (Investigations) | 1
Coagulation time prolonged (Investigations) | 1
Haptoglobin increased (Investigations) | 1
Neutrophil count abnormal (Investigations) | 1
Weight decreased (Investigations) | 4
White blood cell count abnormal (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 12
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Flat affect (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 7
Restlessness (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 3
Urinary retention (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2
Onychalgia (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Embolism (Vascular disorders) | 1
Hot flush (Vascular disorders) | 3
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
On 06 Nov 2012, based on Part I safety findings and due to strategic considerations, Pfizer decided not to open enrolment onto Part II of the study and terminated the study. For primary OM, AEs reported in ≥2 participants overall are presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.